CLINICAL TRIAL: NCT02649075
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Pilot Study Evaluating Serum-Derived Bovine Immunoglobulin / Protein Isolate in the Dietary Management of Mild to Moderate Crohn's Disease
Brief Title: To Evaluate SBI in the Dietary Management of Mild to Moderate Crohn's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: Entera Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EH6112
Record Dates: First submitted 2015-10-12; First posted 2016-01-07 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Crohn's Disease
Keywords: IBD; Inflammatory Bowel Disease; Crohn's; Crohns; SBI; Serum-derived bovine immunoglobulin / protein isolate; EnteraGam
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBI 10 g BID (Active Comparator): Serum-derived Bovine Immunoglobulin / Protein Isolate (SBI) 10.0 grams twice per day
  Interventions: Other: Serum-derived Bovine Immunoglobulin / Protein Isolate
- Placebo BID (Placebo Comparator): Placebo w/control protein
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Serum-derived Bovine Immunoglobulin / Protein Isolate — Serum-derived bovine immunoglobulin protein isolate (SBI) is a specially formulated light-colored protein powder composed of immunoglobulin (IgG) and other serum proteins similar to those found in colostrum and milk. SBI does not contain any milk products such as lactose, casein, or whey. SBI is gluten-free, dye-free, and soy-free. SBI is manufactured in accordance with current Good Manufacturing Practice (cGMP) and FDA guidelines for medical food ingredients. Two packets (each packet contains 5 g of SBI) BID.
  Other Names: EnteraGam
  Arms: SBI 10 g BID
Other: Placebo — Matching placebo with control hydrolyzed gelatin protein. Two packets BID.
  Arms: Placebo BID

SUMMARY:
The objective of this study is to evaluate the nutritional therapy with SBI (a medical food) as compared to placebo in the clinical dietary management of mild to moderate Crohn's disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center, pilot study evaluating SBI 10 g BID compared to matching placebo for 12 weeks followed by a 12 week open-label extension SBI 10 g BID (EnteraGam) in the dietary management of mild to moderate Crohn's disease.

The effect of SBI will be evaluated on Crohn's disease related symptoms and inflammation symptom control as measured by Crohn's disease activity index (CDAI) scores and plasma and stool markers of inflammation. The patient's quality of life will also be assessed as an indicator of disease state.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of mild to moderate Crohn's disease for at least 3 months.
* Screening CDAI between >150 and ≤ 250 based on subject recall.
* Average of greater than two liquid or soft stools per day and an abdominal pain intensity score >1.
* Subject has at least one positive biomarker of inflammation: fecal calprotectin >100 µg/g; elevated C-reactive protein (CRP) >2 mg/dL.

Exclusion Criteria:

* Positive stool test for pathogenic bacteria including Clostridium difficile or O&P.
* Confirmed intestinal stricture with obstructive-like clinical symptoms.
* Bowel resection within the previous 6 months.
* Change in medical therapy: must have been on a stable dose of

  * corticosteroids (prednisone or prednisolone) less than or equal to 20 mg per day for 2 weeks prior to screening,
  * budesonide less than or equal to 9 mg per day for 2 weeks prior to screening,
  * 5-aminosalicylates for 2 weeks prior to screening, and
  * immunomodulators for 6 weeks prior to screening.
* Taking greater than 20 mg per day of a corticosteroid (prednisone or prednisolone) or greater than 9 mg of budesonide.
* Received biologic therapy in past 2 years.
* Diagnosis of one or more co-morbid condition (s) requiring medical or surgical therapy that may affect bowel function, gastrointestinal symptoms.
* Serious infection in the 3 months prior to enrollment.
* Allergy or intolerance to beef or to any ingredient used in the product.
* Participated in an investigational drug or device study within 30 days.
* Does not have access to the internet.
* Taken EnteraGam®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in the number of liquid and soft stools | 12 weeks
Change in abdominal pain intensity score | 12 weeks
Change in fecal calprotectin | 12 weeks
Change in C-reactive protein (CRP) | 12 weeks
Change in Crohn's Disease Activity Index (CDAI) | 12 weeks
Change in plasma albumin levels | 12 weeks
Change in body mass index | 12 weeks
Change in weight | 12 weeks
Change in Quality of Life (SF-36) | 12 weeks

SECONDARY OUTCOMES:
Assess the incidence of adverse events (AEs) and serious AEs (SAEs) | 12 and 24 weeks
Measure clinically significant changes from baseline in vital signs | 12 and 24 weeks
Clinically significant changes from baseline in laboratory testing | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Audrey L Shaw, PhD, Study Director — Entera Health, Inc
Locations (6):
- United States (6):
  - North Little Rock, North Little Rock, Arkansas
  - Hollywood, Hollywood, Florida
  - Winter Park, Winter Park, Florida
  - Hagerstown, Hagerstown, Maryland
  - Manhattan, New York, New York
  - Cincinnati, Cincinnati, Ohio